CLINICAL TRIAL: NCT01361035
Title: Using Effective Provider-Patient Communication to Improve Cancer Screening Among Low Literacy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Eboni Price-Haywood, Adjunct Associate Professor of Clinical Medicine, Tulane University School of Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RWJF-63523
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Cervical Cancer; Breast Cancer; Colorectal Cancer
Keywords: health literacy; cancer screening; doctor-patient communication; standardized patient; continuing medical education
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No communication training (No Intervention): Physicians enrolled in the control arm do not undergo training in health literacy, cancer screening and shared decision making
- Cancer risk ommunication skills training (Other): Physicians enrolled in the intervention arm undergo training in health literacy, cancer screening and shared decision making
  Interventions: Other: Cancer risk communication skills training

INTERVENTIONS:
Other: Cancer risk communication skills training — Intervention physicians receive training in cancer risk communication and shared decision making (SDM). At the end of each visit with intervention physicians, standardized patients (SPs) reveal themselves as actors and give structured verbal feedback. After baseline SP visits, each intervention physician undergoes academic detailing with a communication expert. Intervention physicians are directed to a web-based communication skills tutorial where SP ratings are hyperlinked to key references for supplemental reading. Both study groups will receive annual reports detailing their patients' cancer screening status and aggregate ratings of their communication style.
  Arms: Cancer risk ommunication skills training

SUMMARY:
What's the purpose of this study? This 4-year study is designed: (1) to teach primary care physicians how to recognize low health literacy patients and effectively counsel them on cancer screening using risk communication and shared decision making and (2) to assess the impact of training on changes in physician communication behavior and changes in low health literacy patients' cancer screening behaviors. This study proposal is based on the hypothesis that physician training in cancer screening guidelines, health literacy, and communication skills will improve provider-patient interactions during encounters dealing with preventive health maintenance especially cancer screening.

How will the proposed study be implemented? Thirty-two physicians in the New Orleans metropolitan area will be recruited and randomly assigned to one of two groups. The unit of randomization will be the health care organization or clinic. The intervention group will receive training in health literacy, cancer screening, risk communication and shared decision-making. The control group will not receive communication training until the end of the study. Physicians in both groups will undergo three clinic visits with standardized patients (actors trained to portray real patients; mystery shoppers) but they will not be aware that they are conducting visits with actors. The visits will occur at study enrollment and at 6 and 12 months. At the end of each clinic visit, the standardized patients will rate the physicians' communication skills. Each physician assigned to the intervention group will receive verbal feedback on communication skills from the standardized patients and complete a web-based tutorial. Physicians in the control group will not have access to the web-based tutorial until the end of the study.

For each physician, 10-15 patients with limited health literacy will be recruited to the study. Each patient will rate his/her perceived involvement with care and global satisfaction with care at study enrollment and annually for three years. Age and gender-appropriate referral rates for breast, cervical and colorectal cancer screening and patients' receipt of such screening will be assessed annually for three years. All study physicians, regardless of group assignment, will receive performance feedback (report cards) on their cancer screening rates among low health literacy patients in their clinic.

ELIGIBILITY:
Inclusion Criteria:

Physician

* Physicians who practice at these clinic sites at least one half day per week are eligible to participate in this study.

Patient

* Eligible patients include men and women age 40 to 75, individuals enrolled in the clinic practice for at least one year, and individuals identified as having low or inadequate health literacy via the Rapid Estimate of Adult Literacy in Medicine.

Exclusion Criteria:

Physician

* Any provider planning to leave before the end of 12 months will be excluded.

Patient

* Patients will be excluded if they plan to change primary care provider or site of health plan, have resided in the United States for less than five years, or do not speak English

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in cervical, breast and colorectal cancer screening rates | 0, 12, 24 months
  Cervical/Breast/Colorectal cancer screening rates will be measured at baseline and annually for 2 years to assess whether screening rates improve over time

SECONDARY OUTCOMES:
Change in standardized patient ratings of physician communication behaviors | 0, 6, 12 months
  The mystery shoppers (standardized patients) will rate the physicians' shared decision making and counseling about cancer screening prior to the intervention at baseline and then again at 6-month and 12-month follow up evaluations to assess whether communication behaviors improve over time

CONTACTS AND LOCATIONS:
Overall Officials: Eboni Price-Haywood, MD, MPH, Principal Investigator — Tulane University School of Medicine
Locations (5):
- United States (5):
  - Tulane Communty Health Center at Covenant House, New Orleans, Louisiana
  - Tulane Faculty Practice, New Orleans, Louisiana
  - EXCELth - Ida Hymel Community Health Center, New Orleans, Louisiana
  - DCSNO St Cecelia Medical Center, New Orleans, Louisiana
  - DCSNO Carrollton Medical Center, New Orleans, Louisiana

REFERENCES:
- [Background] Price-Haywood EG, Roth KG, Shelby K, Cooper LA. Cancer risk communication with low health literacy patients: a continuing medical education program. J Gen Intern Med. 2010 May;25 Suppl 2(Suppl 2):S126-9. doi: 10.1007/s11606-009-1211-6. PMID 20352506
- [Result] Price-Haywood EG, Harden-Barrios J, Cooper LA. Comparative effectiveness of audit-feedback versus additional physician communication training to improve cancer screening for patients with limited health literacy. J Gen Intern Med. 2014 Aug;29(8):1113-21. doi: 10.1007/s11606-014-2782-4. Epub 2014 Feb 4. PMID 24590734
- [Derived] Riganti P, Ruiz Yanzi MV, Escobar Liquitay CM, Sgarbossa NJ, Alarcon-Ruiz CA, Kopitowski KS, Franco JV. Shared decision-making for supporting women's decisions about breast cancer screening. Cochrane Database Syst Rev. 2024 May 10;5(5):CD013822. doi: 10.1002/14651858.CD013822.pub2. PMID 38726892